CLINICAL TRIAL: NCT04661228
Title: Diagnosebasert undersøkelse Psykiske Lidelser og Ruslidelser
Brief Title: Diagnostic Survey of Mental and Substance Use Disorders in HUNT (PsykHUNT)
Acronym: PsykHUNT
Status: Completed | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: PDB 2655
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Mental Disorders; Substance Use Disorders; Treatment; Participation
Keywords: Mental Disorders; Substance Use Disorders; Treatment; Participation
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Composite International Diagnostic Interview 5th version (CIDI 5.0) — Observational study assessing prevalence of mental and substance use disorders in the general population

SUMMARY:
The aims of this observational survey are to i) gather experience on how to conduct a prevalence study of mental disorders in the Norwegian setting, ii) collect data on the prevalence, risk factors and consequences of mental and substance use disorders, iii) collect data on treatment coverage for mental and substance use disorders, iv) conduct a thorough nonparticipation analysis.

DETAILED DESCRIPTION:
The psychiatric survey was a sub-project in the fourth wave of the Trøndelag Health Study (HUNT4), conducted on HUNT4 participants aged 20 to 65 years from the geographical areas Nord-Trøndelag and the city of Trondheim. The targeted sample size was 4,000 participants, and 16,602 persons from the study population of HUNT4 participants were invited to reach this goal. The only exclusion criterion was insufficient understanding of Norwegian or English. The investigators had complete lists with postal addresses and mobile phone numbers for all eligible participants as well as information about date of birth and gender. Potential participants were sampled in repeated probability sampling draws over the course of the data-collection period, which lasted from November 2nd 2018 to September 18th 2020. Younger persons were oversampled to adjust for the expected larger nonparticipation among these age-groups. The predesignated participants were informed about the project through postal letters. A week after receipt of the letter, each received an SMS with information on how to sign up for the psychiatric interview. One SMS reminder was sent to persons who did not respond to the initial invitation. The investigators made four contact attempts to schedule the interview amongst those who registered; three by phone and one final by SMS. All participants received a $30 gift card as a token of appreciation. Computer assisted face-to-face or telephone interviews were conducted by trained and certified interviewers at local field stations. The World Health Organization (WHO) Composite International Diagnostic Interview, fifth version (CIDI 5.0) was used as instrument in the data-collection.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of Norwegian or English to conduct the interview

Exclusion Criteria:

* None

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sub-sample of participants from the fourth round of the Trøndelag Health Study (HUNT4). All residents in Trøndelag county of Norway above age 18 were invited to the HUNT4 study.
Sampling Method: Probability Sample
Enrollment: 4242 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of mental and substance use disorders in the general population, and by age, gender, educational attainment and urban/rural residency | November 2018 to September 2020
  Mental and substance use disorders assessed in standardised diagnostic interviews employing the Composite International Diagnostic Interview (CIDI 5.0). Diagnostis criteria after ICD-10 and DSM-V.

SECONDARY OUTCOMES:
The characteristics of nonparticipants in a psychiatric diagnostic survey | November 2018 to September 2020
  Compare characteristics of participants versus nonparticipants in the survey in terms of age, gender, educational attainment, mental health symptoms, alcohol use, and use of health services for mental health problems. Data will be retrieved from the HUNT4 study, and official administrative registries and health registries.
The treatment gap for mental and substance use disorders in the general population | November 2018 to September 2021
  Quantify the gap between perceived need for treatment for mental health problems and received adequate treatment using data from CIDI in linkage with data from official health registries.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reneflot, PhD, Principal Investigator — Norwegian IPH
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Researchers may gain access to participant data by contacting the PsykHUNT publication committee (anne.reneflot@fhi.no). Approval from the Norwegian Regional Committee for Medical and Health Research Ethics (https://helseforskning.etikkom.no) is a pre-requirement. The PsykHUNT dataset is administrated by the HUNT databank. Guidelines for access to PsykHUNT data are found at https://www.ntnu.edu/hunt/data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: June 2021 to September 2030.
Access Criteria: Approval from the Norwegian Regional Committee for Medical and Health Research Ethics (https://helseforskning.etikkom.no). The data must be stored in secure servers which require log in and from which no data can be extracted and copied.

REFERENCES:
- See also: Information in Norwegian about the survey — https://www.fhi.no/cristin-prosjekter/aktiv/diagnosebasert-undersokelse-psykiske-lidelser-og-ruslidelser/